CLINICAL TRIAL: NCT01918319
Title: The Effect of Lifestyle Intervention in Pregnancy - Follow-up on the Offspring in Early Childhood.
Brief Title: Lifestyle in Pregnancy and Offspring
Acronym: LiPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Mette Tanvig, Medical Doctor, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LiPO
Record Dates: First submitted 2013-08-02; First posted 2013-08-07 (Estimated); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Childhood Obesity; Adiposity; Body Composition; Metabolic Risk Factors
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle intervention (Experimental): The active intervention consisted of two major components: dietary counseling and physical activity. Dietary counseling was performed by trained dieticians on four separate occasions at 15, 20, 28 and 35 weeks gestation.
  Interventions: Behavioral: Lifestyle intervention
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Lifestyle intervention — Energy requirements for each participant were individually estimated according to weight and level of activity during pregnancy. Women in the active intervention group were encouraged to be moderately physically active 30-60 minutes a day.Women in this group also had free full time membership in a fitness center for six months. In the fitness centers they had closed training classes with trained physiotherapists for one hour each week.
  Arms: Lifestyle intervention

SUMMARY:
Children born to obese women are at risk of increased adiposity and later adverse metabolic outcomes. We have conducted a follow-up study on an existing clinical trial, called the LiP study (Lifestyle in Pregnancy), registration number NCT00530439,in which 360 obese pregnant women were randomized to either lifestyle intervention or routine obstetric care. This present study follows the children until 3 years of age. We have the hypothesis, that the intervention during pregnancy results in a lower degree of adiposity and metabolic risk factors in the offspring. Clinical examination is taking place at age 2.5-3 years including anthropometric measurements, Dual energy x-ray (DXA) scans and blood samples measuring metabolic markers.

ELIGIBILITY:
Inclusion Criteria:

* children born to women who were part of the preceding LiP study and who completed the LiP study until birth. Inclusion criteria for the LiP study:
* singleton pregnant
* BMI >/= 30 and </= 45 E xclusion Criteria for preceding LiP study:
* Chronic diseases
* Not Danish speaking
* Abuse of alcohol or drugs
* Preterm delivery in earlier pregnancies

Ages: 30 Months to 40 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 157 (Actual)
Dates: Start 2011-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Body Mass Index standard deviation score | On average 2.9 years of age

SECONDARY OUTCOMES:
Fat mass percent | On average 2.9 years of age
  Fat mass estimated by dxa scans.

OTHER OUTCOMES:
Anthropometric and metabolic risk factors and bone mineralization | On average 2.9 years of age
  BMI, Skinfold thicknesses, abdominal circumference, hip circumference, abdominal to hip circumference ratio, height, weight. DXA scan: fat mass, fat mass percent, lean mass, lean mass percent, body fat distribution. Bone mass density, bone mass content. Fasting blood glucose, HbA1C, fasting insulin, fasting c-peptide, fasting lipids; HDL; LDL, triglycerides, total cholesterol. 25-hydroxy vitamin D. Bone mineralization measured by dual energy x-ray

CONTACTS AND LOCATIONS:
Overall Officials: Mette Tanvig, MD, Principal Investigator — Department of endocrinology, Odense University Hospital
Locations (1):
- Department of Endocrinology, Odense University Hospital, Odense, Denmark

REFERENCES:
- [Background] Vinter CA, Jensen DM, Ovesen P, Beck-Nielsen H, Jorgensen JS. The LiP (Lifestyle in Pregnancy) study: a randomized controlled trial of lifestyle intervention in 360 obese pregnant women. Diabetes Care. 2011 Dec;34(12):2502-7. doi: 10.2337/dc11-1150. Epub 2011 Oct 4. PMID 21972411
- [Derived] Luef BM, Stentebjerg LL, Tanvig MH, Aalders J, Moller S, Ovesen PG, Christesen HT, McIntyre HD, Catalano PM, Jorgensen JS, Overgaard M, Jensen DM, Vinter CA. Impact of maternal fasting blood glucose in pregnancy on body composition, anthropometric, and metabolic outcomes in newborns and 3-Year-Old offspring: results from the lifestyle in pregnancy and offspring study. BMC Pregnancy Childbirth. 2026 Jan 29. doi: 10.1186/s12884-026-08692-3. Online ahead of print. PMID 41612293
- [Derived] Tanvig M, Vinter CA, Jorgensen JS, Wehberg S, Ovesen PG, Beck-Nielsen H, Christesen HT, Jensen DM. Effects of lifestyle intervention in pregnancy and anthropometrics at birth on offspring metabolic profile at 2.8 years: results from the Lifestyle in Pregnancy and Offspring (LiPO) study. J Clin Endocrinol Metab. 2015 Jan;100(1):175-83. doi: 10.1210/jc.2014-2675. PMID 25343235
- [Derived] Tanvig M, Vinter CA, Jorgensen JS, Wehberg S, Ovesen PG, Lamont RF, Beck-Nielsen H, Christesen HT, Jensen DM. Anthropometrics and body composition by dual energy X-ray in children of obese women: a follow-up of a randomized controlled trial (the Lifestyle in Pregnancy and Offspring [LiPO] study). PLoS One. 2014 Feb 24;9(2):e89590. doi: 10.1371/journal.pone.0089590. eCollection 2014. PMID 24586896